CLINICAL TRIAL: NCT03602469
Title: Efficacy of Magnesium Sulfate Added to Bupivacaine in Suprascapular Nerve Block on Duration of Analgesia Following Shoulder Arthroscopy: a Prospective Randomized Controlled Study
Brief Title: Postoperative Analgesia of Magnesium Sulfate in Suprascapular Nerve Block Following Shoulder Arthroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R ∕18.04.172
Record Dates: First submitted 2018-06-20; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-06

CONDITIONS: Arthroscopic Shoulder Surgery
MeSH Terms: interventions — Bupivacaine; Propofol; Ultrasonography; Sevoflurane; Rocuronium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine (Experimental): Ultrasound-guided suprascapular nerve block using bupivacaine will be performed before induction of general anesthesia
  Interventions: Drug: Bupivacaine; Drug: Propofol; Device: Ultrasound; Drug: Sevoflurane; Drug: Rocuronium
- Bupivacaine-magnesium (Active Comparator): Ultrasound-guided suprascapular nerve block using bupivacaine in conjunction of magnesium sulfate will be performed before induction of general anesthesia
  Interventions: Drug: Bupivacaine-magnesium; Drug: Propofol; Device: Ultrasound; Drug: Sevoflurane; Drug: Rocuronium

INTERVENTIONS:
Drug: Bupivacaine — Ultrasound-guided suprascapular nerve block will be performed using 7 mL of 0.5% bupivacaine plus 3 mL of 0.9% saline
  Arms: Bupivacaine
Drug: Bupivacaine-magnesium — Ultrasound-guided suprascapular nerve block will be performed using 7 mL of 0.5% bupivacaine plus magnesium sulfate 10% (3 ml) (total 10mL)
  Arms: Bupivacaine-magnesium
Drug: Propofol — Using propofol 1.5-2.5 mg/kg
Device: Ultrasound — Ultrasound-guided suprascapular nerve block
Drug: Sevoflurane — Sevoflurane 0.7-1.5 MAC in 40% oxygen
Drug: Rocuronium — Rocuronium 0.6 mg/kg

SUMMARY:
* Arthroscopic shoulder surgeries in adults are accompanied with severe immediate postoperative pain reported in approximately 45% of patients. For quicker recovery and rehabilitation of these patients, postoperative analgesia is mandatory.
* Different analgesic modalities have been proposed including parenteral opioids, intra-articular injection of local anesthetics, interscalene brachial plexus block (ISB), and a suprascapular nerve block (SSNB), with varying degrees of effectiveness and multiple reported side effects.
* A recent meta-analysis demonstrates that suprascapular block results in 24-h morphine consumption and pain scores similar to ISB, so, it may be considered an effective and safe alternative for interscalene block in shoulder surgery, with less motor restriction, and fewer complications.
* Different agents are used as adjuvants to local anesthetics during peripheral nerve block to prolong its analgesic action including magnesium sulfate.
* A meta-analysis by Mengzhu et al., concluded that magnesium sulfate combined with local anesthetics in perineural nerve blocks provided better analgesic efficacy and may be a promising analgesic for perineural nerve blocks.
* Antinociceptive effects of magnesium are due to the regulation of calcium influx into the cell and a non-competitive antagonism of the NMDA receptors

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effects of magnesium sulfate as an adjuvant to bupivacaine in suprascapular nerve block on the duration and quality of postoperative analgesia following shoulder arthroscopy, postoperative pain VAS scores, intraoperative fentanyl requirements, sedation scores, respiratory depression, postoperative 24 hours cumulative morphine consumption.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-III

Exclusion Criteria:

* Patient's refusal
* Significant cardiac diseases
* Significant hepatic diseases
* Significant renal diseases (serum creatinine ˃ 1.5 mg/dl)
* Cardiac conduction abnormalities
* Drug abuse
* Pregnancy
* Allergy to study medications
* Mental disease
* Communication barrier
* Coagulopathy
* Local skin infection
* Traumatic nerve injury of upper limb
* Patients receiving opioid analgesics
* Patients receiving magnesium sulfate
* Patients receiving beta blockers
* Patients receiving calcium channel blockers
* Previous shoulder surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Duration of postoperative analgesia | For 8 hours after suprascapular nerve block
  time from administering the study solution in the suprascapular block till the time for the first rescue morphine request

SECONDARY OUTCOMES:
Pain score at rest | time 0 (after extubating) and at 30 minutes, 1 hour , 2 hours, 4hours, 6hours, 8hours,12 hours , 16hours, 20 hours and 24 hours postoperatively
  Pain score as assessed using visual analogue scale to assess the severity of postoperative pain (0 mm for no pain and 100 mm for worst imaginable pain)
Pain score on shoulder abduction | time 0 (after extubating) and at 30 minutes, 1 hour , 2 hours, 4hours, 6hours, 8hours,12 hours , 16hours, 20 hours and 24 hours postoperatively
  Pain score as assessed using visual analogue scale to assess the severity of postoperative pain (0 mm for no pain and 100 mm for worst imaginable pain)
Systolic arterial blood pressure | At baseline, immediately after induction of anaesthesia, at skin incision, every 15 minutes till the end of surgery, on arrival to PACU, then at 30, 60 minutes after surgery , every 6 hours up to 24 hours postoperatively
Diastolic arterial blood pressure | At baseline, immediately after induction of anaesthesia, at skin incision, every 15 minutes till the end of surgery, on arrival to PACU, then at 30, 60 minutes after surgery , every 6 hours up to 24 hours postoperatively
Heart rate | At baseline, immediately after induction of anaesthesia, at skin incision, every 15 minutes till the end of surgery, on arrival to PACU, then at 30, 60 minutes after surgery ,every 6 hours up to 24 hours postoperatively
Intraoperative fentanyl requirements | For 5 hours after suprascapular nerve block
Sedation scores | at 1 hour, 2 hours, and 6 hours postoperatively
  Sedation: will be assessed using a sedation scale (awake and alert= 0; quietly awake= 1; asleep but easily roused= 2; deep asleep= 3).
The degree of nausea and vomiting | For 24 hours after surgery
  Nausea will be measured using a numerical rating system (none= 0; mild= 1; moderate= 2; severe= 3)
Number of vomiting episodes | For 24 hours after surgery
Number of antiemetics received | For 24 hours after surgery
Postoperative cumulative morphine consumption | For 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hanaa M Elbendary, MD, Study Chair — Assistant Professor, MD anesthesia Department, Faculty of Medicine, Mansoura University, Egypt
Locations (1):
- Mansoura University, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided